CLINICAL TRIAL: NCT02461563
Title: A Multiple-Dose Study to Evaluate the Safety, Pharmacodynamics and Pharmacokinetics of MK-1075 in GT3 and GT1 HCV Infected Patients
Brief Title: A Multiple-Dose Study to Evaluate MK-1075 in Hepatitis C Virus (HCV) Infected Participants (MK-1075-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1075-004; 2015-001687-18 (EudraCT Number)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- GT1: 200 mg MK-1075 (Experimental): Fasted GT1 participants are administered 200 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
  Interventions: Drug: 200 mg MK-1075
- GT1: 400 mg MK-1075 (Experimental): Fasted GT1 participants are administered 400 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
  Interventions: Drug: 400 mg MK-1075
- GT1: 800 mg MK-1075 (Experimental): Fasted GT1 participants are administered 800 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
  Interventions: Drug: 800 mg MK-1075
- GT3: 200 mg MK-1075 (Experimental): Fasted GT3 participants are administered 200 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
  Interventions: Drug: 200 mg MK-1075
- GT3: 400 mg MK-1075 (Experimental): Fasted GT3 participants are administered 400 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
  Interventions: Drug: 400 mg MK-1075
- GT3: 800 mg MK-1075 (Experimental): Fasted GT3 participants are administered 800 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
  Interventions: Drug: 800 mg MK-1075

INTERVENTIONS:
Drug: 200 mg MK-1075 — Two 100 mg tablets of MK-1075 administered orally, once daily for 7 consecutive days
  Arms: GT1: 200 mg MK-1075; GT3: 200 mg MK-1075
Drug: 400 mg MK-1075 — Four 100 mg tablets of MK-1075 administered orally, once daily for 7 consecutive days
  Arms: GT1: 400 mg MK-1075; GT3: 400 mg MK-1075
Drug: 800 mg MK-1075 — Eight 100 mg tablets of MK-1075 administered orally, once daily for 7 consecutive days
  Arms: GT1: 800 mg MK-1075; GT3: 800 mg MK-1075

SUMMARY:
This study will evaluate safety, pharmacokinetics (PK), and the ability of MK-1075 to suppress viral load (VL) in HCV-infected participants during 7 days of once daily dose administration. The primary hypothesis is at a once-daily dose that is sufficiently safe and well tolerated in HCV-infected participants, the mean maximum HCV RNA (log10 IU/mL) reduction is at least 3 log10 IU/mL as compared to baseline following multiple dose oral administration of MK-1075 in HCV genotype 1 (GT1) and genotype 3 (GT3) infected participants.

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential
* Have a body mass index (BMI) >=18 to =< 37 kg/m^2
* Excepting HCV infection, be in good health
* Have a clinical diagnosis of chronic HCV infection, exclusively GT1 or exclusively GT3
* Agree to follow smoking restrictions

Exclusion Criteria:

* Has a history of clinically significant, not stably controlled endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or diseases.
* Have been treated with amiodarone within the prior year, or is currently on beta-blockers or verapamil
* Has a history of cancer (malignancy)
* Has a history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Is positive for hepatitis B surface antigen or human immunodeficiency virus (HIV)
* Has had major surgery, donated or lost approximately 500 mL blood within 4 weeks prior to screening visit
* Has participated in another drug trial within 4 weeks prior to screening visit
* Is taking a non-permitted medication to treat a co-morbid condition
* Consumes greater than 2 glasses of alcoholic beverages
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 12 months
* Has evidence or history of chronic hepatitis not caused by HCV, including but not limited to non-HCV viral hepatitis, non-alcoholic steatohepatitis (NASH), drug-induced hepatitis, or autoimmune hepatitis
* Has been treated with other HCV inhibitors, such as sofosbuvir or VX-135
* Has evidence of advanced or decompensated liver disease, bridging fibrosis or higher grade fibrosis from a prior liver biopsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males or females of non-child bearing potential with verified Genotype 1 (GT1) or Genotype 3 (GT3) Hepatitis C Virus (HCV) infection, between the ages of 18 and 65 years (inclusive) were enrolled in this trial.
Pre-assignment Details: GT1 and GT3 participants planned to receive 200 mg MK-1075 were not treated based on available data from previous studies.
Groups:
- GT1 400 mg MK-1075: Fasted GT1 participants were administered 400 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
- GT1 MK-1075 600 mg: Fasted GT1 participants were administered 600 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
- GT3 400 mg MK-1075: Fasted GT3 participants were administered 400 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
- GT3 600 mg MK-1075: Fasted GT3 participants were administered 600 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
Period: Overall Study
Arm/Group | GT1 400 mg MK-1075 | GT1 MK-1075 600 mg | GT3 400 mg MK-1075 | GT3 600 mg MK-1075
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GT1 400 mg MK-1075 | GT1 MK-1075 600 mg | GT3 400 mg MK-1075 | GT3 600 mg MK-1075 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (9.3) | 39.7 (11.0) | 39.0 (3.0) | 46.0 (7.0) | 41.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2
  Male | 3 | 3 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Day 42
Population: Participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | GT1 400 mg MK-1075 | GT1 MK-1075 600 mg | GT3 400 mg MK-1075 | GT3 600 mg MK-1075
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 3 | 2 | 3 | 2

2. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 1
Time Frame: Up to Day 7
Population: Participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | GT1 400 mg MK-1075 | GT1 MK-1075 600 mg | GT3 400 mg MK-1075 | GT3 600 mg MK-1075
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Change From Baseline in Maximum log10 HCV RNA Following Multiple Dose Oral Administration of MK-1075
Description: Blood was collected on Days 1, 3, 4, 5, 6, 7, 21, 28 and 42, where baseline measurement was defined as the measurement obtained pre-dose on the first day of dosing. Change from baseline in log10 HCV RNA levels, was determined, and the maximum reduction in HCV RNA was analyzed by an ANOVA model with a fixed effect for treatment. The primary hypothesis is, with a posterior probability larger than 70%, there is at least a 3 log10 reduction from baseline in HCV RNA.
Time Frame: Day 1 (pre-dose, 2, 4, 8, 12, and 24 hours postdose); Days 3, 4, 5, 6 (pre-dose); Day 7 (predose, 4, 12, 24, 48, 72, 96, 120, and 192 hours postdose); Days 21, 28 and 42
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements and absence of major protocol deviations.
Measure: Least Squares Mean (90% Confidence Interval); unit: log10 IU/mL
Arm/Group | GT1 400 mg MK-1075 | GT1 MK-1075 600 mg | GT3 400 mg MK-1075 | GT3 600 mg MK-1075
Number analyzed (Participants) | 3 | 3 | 3 | 3
log10 IU/mL | 3.465 [2.427 to 4.502] | 4.122 [3.084 to 5.159] | 4.071 [3.034 to 5.109] | 5.132 [4.095 to 6.169]

4. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to 24 Hrs (AUC 0-24hr) of MK-1075 Following Multiple Dose Oral Administration of MK-1075
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma AUC 0-24hr of MK-1075 for pooled GT1 and GT3 genotypes. A non-compartmental analysis on MK-1075 plasma concentrations was performed where actual sampling times, converted to elapsed time relative to dosing times, by using the software Phoenix WinNonlin® Professional (Version 6.3). AUC was calculated using the linear-up/log-down trapezoidal method.
Time Frame: Day 7 at the following time points: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: AUC 0-24hr were not determined because concentrations of MK-1075 at 24 hour were not quantifiable
Groups:
- GT1 and GT3 Pooled 400 mg MK-1075: Fasted GT1 and GT3 participants were administered 400 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
- GT1 and GT3 Pooled MK-1075 600 mg: Fasted GT1 and GT3 participants were administered 600 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
Arm/Group | GT1 and GT3 Pooled 400 mg MK-1075 | GT1 and GT3 Pooled MK-1075 600 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: AUC 0-24hr of Metabolite M1 Following Multiple Dose Oral Administration of MK-1075
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma AUC 0-24hr of the MK-1075 metabolite M1 for pooled GT1 and GT3 genotypes. A non-compartmental analysis on M1 plasma concentrations was performed where actual sampling times, converted to elapsed time relative to dosing times, by using the software Phoenix WinNonlin® Professional (Version 6.3). AUC was calculated using the linear-up/log-down trapezoidal method.
Time Frame: Day 7 at the following time points: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μmol/L
Arm/Group | GT1 and GT3 Pooled 400 mg MK-1075 | GT1 and GT3 Pooled MK-1075 600 mg
Number analyzed (Participants) | 6 | 6
hr*μmol/L | 35.3 (12.9) | 51.2 (12)

6. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to Last (AUC 0-last) of MK-1075 Following Multiple Dose Oral Administration of MK-1075
Description: Blood was collected from pre-dose up to 120 hours post-dose in order to determine the plasma AUC 0-last of MK-1075 for pooled GT1 and GT3 genotypes. A non-compartmental analysis on MK-1075 plasma concentrations was performed where actual sampling times, converted to elapsed time relative to dosing times, by using the software Phoenix WinNonlin® Professional (Version 6.3). AUC was calculated using the linear-up/log-down trapezoidal method.
Time Frame: Day 7 at the following time points: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μmol/L
Arm/Group | GT1 and GT3 Pooled 400 mg MK-1075 | GT1 and GT3 Pooled MK-1075 600 mg
Number analyzed (Participants) | 6 | 6
hr*μmol/L | 1.1 (41.3) | 0.89 (54.2)

7. Secondary Outcome: AUC 0-last of Metabolite M1 Following Multiple Dose Oral Administration of MK-1075
Description: Blood was collected from pre-dose up to 120 hours post-dose in order to determine the plasma AUC 0-last of M1 for pooled GT1 and GT3 genotypes. A non-compartmental analysis on M1 plasma concentrations was performed where actual sampling times, converted to elapsed time relative to dosing times, by using the software Phoenix WinNonlin® Professional (Version 6.3). AUC was calculated using the linear-up/log-down trapezoidal method.
Time Frame: Day 7 at the following time points: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μmol/L
Arm/Group | GT1 and GT3 Pooled 400 mg MK-1075 | GT1 and GT3 Pooled MK-1075 600 mg
Number analyzed (Participants) | 6 | 6
hr*μmol/L | 62.2 (29.6) | 90.6 (20.9)

8. Secondary Outcome: Plasma Concentration at 24 Hours Post-dose (C24hr) of MK-1075 Following Multiple Dose Oral Administration of MK-1075
Description: Blood was collected at 24 hours post-dose in order to determine the plasma C24hr of MK- 1075 for pooled GT1 and GT3 genotypes. A non-compartmental analysis on MK-1075 plasma concentrations was performed where actual sampling times, converted to elapsed time relative to dosing times, by using the software Phoenix WinNonlin® Professional (Version 6.3).
Time Frame: Day 7 at 24 hours postdose
Population: C24hr were not determined because concentrations of MK-1075 at 24 hour were not quantifiable.
Arm/Group | GT1 and GT3 Pooled 400 mg MK-1075 | GT1 and GT3 Pooled MK-1075 600 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: C24hr of Metabolite M1 Following Multiple Dose Oral Administration of MK-1075
Description: Blood was collected at 24 hours post-dose in order to determine the plasma C24hr of MK-1075 metabolite M1 for pooled GT1 and GT3 genotypes. A non-compartmental analysis on M1 plasma concentrations was performed where actual sampling times, converted to elapsed time relative to dosing times, by using the software Phoenix WinNonlin® Professional (Version 6.3).
Time Frame: Day 7 at 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/L
Arm/Group | GT1 and GT3 Pooled 400 mg MK-1075 | GT1 and GT3 Pooled MK-1075 600 mg
Number analyzed (Participants) | 6 | 6
μmol/L | 0.561 (39.9) | 0.947 (25.8)

ADVERSE EVENTS:
Time Frame: Pre-treatment: 28 days before treatment up to Treatment; Treatment: Day 1 up to Day 7; Post-Treatment: Day 8 up to day 42
Description: Participants who received at least one dose of the investigational drug. Adverse events are also reported for GT1 and GT3 arms during Pre-treatment and Post-study periods.
Groups:
- GT1 Pre-treatment: GT1 participants were enrolled for 4 weeks prior to randomization and treatment.
- GT3 Pre-treatment: GT3 participants were enrolled for 4 weeks prior to randomization and treatment.
- GT1 600 mg MK-1075: Fasted GT1 participants were administered 600 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days
- GT3 MK-1075 400 mg: Fasted GT3 participants were administered 400 mg MK-1075 in tablet form, orally, once daily for 7 consecutive days.
- GT1 Post-study: After treatment Day 7, GT1 participants were monitored for AEs up to Day 42.
- GT3 Post-study: After treatment Day 7, GT3 participants were monitored for AEs up to Day 42.
Arm/Group | GT1 Pre-treatment | GT3 Pre-treatment | GT1 400 mg MK-1075 | GT1 600 mg MK-1075 | GT3 MK-1075 400 mg | GT3 600 mg MK-1075 | GT1 Post-study | GT3 Post-study
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 3/3 | 2/3 | 3/3 | 2/3 | 1/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GT1 Pre-treatment (N=6) | GT3 Pre-treatment (N=6) | GT1 400 mg MK-1075 (N=3) | GT1 600 mg MK-1075 (N=3) | GT3 MK-1075 400 mg (N=3) | GT3 600 mg MK-1075 (N=3) | GT1 Post-study (N=6) | GT3 Post-study (N=6)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.